CLINICAL TRIAL: NCT06587633
Title: 3D BIO-STRUCTURES POPULATED WITH MICRO-FRAGMENTED, EMULSIFIED STROMAL TISSUE DERIVED FROM AUTOLOGOUS ADIPOSE TISSUE HARVESTING FOR THE REGENERATIVE TREATMENT OF POST-SURGICAL DEFECTS OF THE GASTROINTESTINAL TRACT
Brief Title: 3D BIO-STRUCTURES FOR G.I. POST-SURGICAL DEFECTS
Acronym: 3DReG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: IRCCS Ospedale Casa Sollievo della Sofferenza (Unknown)
Responsible Party: Principal Investigator, Papi Massimiliano, professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6913
Record Dates: First submitted 2024-08-28; First posted 2024-09-19 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Fistula
MeSH Terms: conditions — Fistula | interventions — Endoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic procedure (Experimental)
  Interventions: Device: Endoscopic procedure

INTERVENTIONS:
Device: Endoscopic procedure — tSVFem injection + 3D scaffold placement

SUMMARY:
The study is focused on evaluating the safety and efficacy of using vascular stromal tissue, derived from autologous adipose tissue, and subjected to microfragmentation and emulsification (Stromal Vascular Fraction Micro-Emulsion - tSVFem), in the treatment of chronic gastrointestinal fistulae (CGF). Tissue regeneration will be stimulated using 3D bio-printed scaffolds, enriched at implantation with mesenchymal stem cells derived from patients' adipose tissue; injection of tSVFem and scaffold placement will be performed endoscopically. The study proposes to use 3D bioprinting to create customized polymeric bioinks (gels) on supporting scaffolds that can serve as a framework for the growth and development of the patient's cells. This approach aims to promote tissue regeneration and integration, repair extensive CGF and restore the proper microbiota.

A small portion of the patient's tSVFem will be injected in a bioreactor into the scaffolds and used for evaluation of the ability of the scaffolds to support cell proliferation, migration, and differentiation, as well as secretion of cytokines and growth factors and the immunological response. Also, to analyze the effect on cells and microbial species, the intestinal microbiota will be analyzed in a bioreactor under different dynamic conditions on the growth and differentiation of the MSCs contained in tsVFem, on the bio-printed scaffolds and the immunological results.

ELIGIBILITY:
Inclusion Criteria:

* patients with CGF at any level that can be approached endoscopically and for whom the possibility of conventional conservative treatment is ruled out, or all possible conservative or surgical treatments have already been performed without benefit, or in whom the reiteration of such treatments is contraindicated, because of life-threatening, and/or possible complications, and/or disabling outcomes.

Exclusion Criteria:

* patients who have not given informed consent to the procedure;
* patients with entero-enteral CGF,
* patients who have therapeutic options of other type.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-06-10 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the custom-made 3D printed vascular stromal tissue and scaffolds to treat CGFs. | 24 months
  Efficacy: endoscopic evaluation with or without radiological auxilium at 3 months after the procedure. Fistula will be described as: closed or still open. Further endoscopic evaluations with or without radiological auxilium could be repeated to assess maintenance of the closure.

SECONDARY OUTCOMES:
Evaluation of immunological response | 24 months
  Exposure of the tSVFem-containing scaffolds to peripheral blood mononuclear cells obtained from the same patient. Microbiota analysis (obtained from stool sample of the patient) before and after the treatment. DNA extraction, metagenomics or 16S rRNA gene sequencing will be used to determine the diversity and abundance of the microbial community. Statistical analysis will be performed to identify specific microbial taxa that have changed significantly. PICRUSt2 and ALDEx2 tools will be applied to identify microbial signatures
Incidence of Treatment-Emergent Adverse Events | 24 months
  treatment-related adverse events as assessed by CTCAE v5.0 will be registered during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino gemelli IRCCS, Roma, Italy